CLINICAL TRIAL: NCT06154330
Title: Safety and Efficacy of Suprachoroidal Tube Shunt in Patients With Primary Open and Pseudoexfoliation Glaucomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Davinci LTD (Other)
Responsible Party: Principal Investigator, Nikoloz Labauri, Founder and Managing Director, Principal Investigator, Davinci LTD
Other Study IDs: SCS_001
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma, Open-Angle; Suprachoroidal Space; Pseudo Exfoliation Syndrome
Keywords: MIGS; Suprachoroidal Space; Glaucoma, Open-Angle; Suprachoroidal Silicone Tube; Suprachoroidal Shunt; Glaucoma Shunt
MeSH Terms: conditions — Glaucoma, Open-Angle; Choroidal Effusions; Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess safety and efficacy of a novel suprachoroidal silicone tube (SST) shunt for the treatment of primary open angle and exfoliative glaucomas.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects from 40 years up to 90 years old
* Diagnosis of primary open angle glaucoma (POAG) and pseudo-exfoliative glaucoma
* Subject is able to understand and sign a written informed consent form
* Subject who underwent SST implantation and agreed to come for the cross-sectional follow-up

Exclusion Criteria:

* Close angle forms of glaucoma
* Congenital or developmental glaucoma
* Pseudophakic with an anterior chamber intraocular lens (IOL), iris fixed IOL, or implantable contact lens (ICL)
* Prior glaucoma procedures such as Selective Laser Trabeculoplasty (SLT), Microinvasive Glaucoma Surgery (MIGS) or Episcleral Shunts
* History of corneal transplant, corneal refractive surgery, corneal dystrophy, or corneal ectasia (such as either keratoconus or keratoglobus) in the study eye
* Chronic ocular inflammatory disease, or clinically significant ocular inflammation or infection (e.g., uveitis, iritis, iridocyclitis, retinitis).
* Any condition that, in the Investigator´s opinion, can interfere with full participation in the study, including study treatment and attending required visits; can pose a significant risk to the participant, or interfere with interpretation of study data.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All study patients were Caucasian
Sampling Method: Non-Probability Sample
Enrollment: 91 (Estimated)
Dates: Start 2023-11-20 (Actual); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-23 (Estimated)

PRIMARY OUTCOMES:
Main outcome measures | 1 month
  A successful outcome was defined as Intraocular Pressure (IOP) reduction in ≥20%, with the IOP range 5-21mm/Hg. Successful outcomes were further categorized into two groups: Complete success - IOP reduction in ≥20%, with unmedicated the IOP range 5-21mm/Hg and Qualified success where reduction and ranges of IOP is the same but with antiglaucoma medications. Failure was defined as IOP reduction in <20% or IOP >21mm/Hg at last follow up. Permanent hypotony was defined as IOP < 5mm/Hg during more than 4 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Davinci Eye Center, LTD, Tbilisi, Georgia

IPD SHARING:
Plan to Share IPD: Undecided